CLINICAL TRIAL: NCT00533845
Title: Intraperitoneal Bupivicaine Infusion Using the On-Q Pain Pump After Laparoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Danny A Sherwinter, Attending, Surgery, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07/02/VA13
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-Q pain pump (Experimental): Bupivacaine
  Interventions: Drug: On-Q Pain Pump
- Placebo/control (Placebo Comparator): Saline
  Interventions: Drug: On-Q Pain Pump

INTERVENTIONS:
Drug: On-Q Pain Pump — Bupivicaine .375% via on-Q pump will be infused at a rate of 2cc/hr intraperitoneally
  Other Names: Marcaine

SUMMARY:
After Laparoscopic surgery most patients experience some form of mild to moderate pain. The current standard of care is to treat this pain with local anesthetics (numbing medication, that deadens the nerve endings) to the small surgical incisions (cuts) and narcotic systemic analgesics (medication injected into your vein to control pain such as morphine).

Although this treatment improves pain symptoms it is not perfect. Firstly, complete pain control is rarely achieved and secondly, narcotics (such as morphine) often have many side effects including nausea, vomiting, sedation (sleepiness), constipation and abdominal upset. All of these issues make recovery less comfortable and delays return to full function (work, school and other activities of daily life).

A new FDA approved device is now available that offers the benefits of long term anesthesia without the side effects of narcotics. It consists of a pump that continuously infuses local anesthesia into and around the surgical site. This pump is placed during your operation. You then carry a tennis ball sized container made of soft plastic in a pouch which drips numbing medicine around your wounds for 2 days continuously.

The purpose of this study is to see if this pump improves postoperative pain, decreases the need for narcotic pain medicine and allows people to return to their activities earlier.

DETAILED DESCRIPTION:
The procedure of the current study is to randomly assign patients undergoing minimally invasive surgeries (laparoscopic cholecystectomies and laparoscopic Lap-Banding procedures) to one of two groups. Both groups will have the standard surgical procedure performed and then at the completion will have the on-Q system placed in a subdiaphragmatic (within the abdomen) location. Half of the study group will have bupivicaine, a numbing medicine in the pump while the other half will have sterile saline in their pump. Neither the patient nor the surgeon will be aware of which group any particular patient is in, this is a process known as "blinding" and improves the reliability of the results. All patients will receive the standard locally infiltrated trocar site local anesthetic and either a prescription for Vicodin for ambulatory patients or morphine injected into their vein for patients staying in the hospital.

All patients will then be asked at preset intervals their level of pain the presence of nausea and their need for Vicodin or morphine. Ambulatory patients will be reached by phone for answers to these questions. All patients will have their pain controlled in the usual and standard way at all times. The On-Q pump will be removed at 48hours.

The results will then be statistically reviewed to see if the On-Q pumps were of benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy or Lap-Band ASA III or less

Exclusion Criteria:

* Patients who refuse consent
* Are converted from laparoscopy to open surgery
* Are allergic to bupivacaine
* Are unable to followup

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny A Sherwinter, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 participant randomized to bupivicaine did not complete the study because the participant had to be returned to surgery prior to commencement of study procedures
Groups:
- Bupivacaine: On-Q pump containing Bupivacaine implanted
  On-Q Pain Pump: Bupivicaine .375% via on-Q pump will be infused at a rate of 2cc/hr intraperitoneally
- Placebo/Control: Saline used in the implanted On-Q device
Period: Overall Study
Arm/Group | Bupivacaine | Placebo/Control
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis - 30 enrolled but only 29 evaluated because patient required re-operative intervention with removal of experimental device precluding assessment of VAS pain scores
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Placebo/Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (9.7) | 42.0 (11.8) | 43.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 4 | 4 | 8
Pain Scale [Mean (Standard Deviation); unit: units on a scale] — Likert scale ranging from 0 to 10 (0 being no pain and 10 being very severe pain)
  units on a scale | 3.5 (.75) | 3.5 (.75) | 3.5 (.75)

OUTCOME MEASURES:

1. Primary Outcome: Visual Aanalog Scale (VAS) for Pain Assessment With Cough at 48 Hours
Description: Pain assessment using a subjective pain visual analog scale VAS with cough at 48 hours. Participant will be shown a card that has a visual analogue (Faces) pains scale combined with numerical (0-10) analogue scale (0 is no pain, 10 is the worst pain imaginable).
Time Frame: 48 hours postop
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine | Placebo/Control
Number analyzed (Participants) | 14 | 15
units on a scale | 1.7 (1.94) | 3.9 (2.88)
Statistical Analysis 1: Comparison: Bupivacaine vs Placebo/Control; Test type: Superiority or Other; p = .0022, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Bupivacaine | Placebo/Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No